CLINICAL TRIAL: NCT05077124
Title: Safe and Timely Antithrombotic Removal (STAR) Registry: International Registry on the Use of CytoSorb for Removal of Antithrombotic Agents in the Acute Hospital Setting
Brief Title: Safe and Timely Antithrombotic Removal (STAR) Registry
Status: Recruiting | Type: Observational
Sponsor: CytoSorbents, Inc (Industry)
Responsible Party: Sponsor
Other Study IDs: O05
Record Dates: First submitted 2021-09-09; First posted 2021-10-14 (Actual); Last update posted 2025-07-16 (Actual); Status verified 2025-07

CONDITIONS: Hemorrhage, Surgical; Hemorrhage Postoperative; Blood Loss, Surgical; Blood Loss, Postoperative
MeSH Terms: conditions — Blood Loss, Surgical; Postoperative Hemorrhage

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Device: CytoSorb — Sorbent hemoperfusion system

SUMMARY:
This registry will capture real-world clinical use patterns and associated clinical outcomes with the use of CytoSorb for the removal of antithrombotic agents.

DETAILED DESCRIPTION:
The STAR Registry will collect patient-level clinical data on antithrombotic removal with CytoSorb. The decision to use CytoSorb in this clinical setting is based on the clinical rationale of mitigating the high risk of bleeding events that is directly linked to the presence of the antithrombotic agent. This registry is to capture real-world clinical use patterns and associated clinical outcomes with the use of CytoSorb. Data of retrospective and prospective patients will be included in the registry. Safety will be assessed by collection of (at least possibly) device-related adverse events. Data collection is done up to 30 days post-operation.

ELIGIBILITY:
Inclusion Criteria:

* CytoSorb utilization for antithrombotic removal
* Informed consent for prospective registry participation

Exclusion Criteria:

• Use of CytoSorb for purpose other than antithrombotic removal

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients undergoing invasive management, including surgery, who receive CytoSorb therapy for antithrombotic removal as part of their routine clinical care can be included in this registry
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2021-09-30 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
Bleeding complications including requirements for transfusions and other blood products | Assessed until postoperative day (POD) 3, date of ICU discharge, or date of death, whatever comes first; on average 3 days

CONTACTS AND LOCATIONS:
Overall Officials: Michael Schmoeckel, Prof, MD, Principal Investigator — LMU Klinikum Großhadern; Robert Storey, Prof, BSc, Principal Investigator — University of Sheffield
Locations (30):
- Austria (4):
  - Universitätsklinikum Graz, Graz
  - Medizinische Universität Innsbruck, Innsbruck
  - Klinikum Klagenfurt am Wörthersee, Klagenfurt
  - Medical University of Vienna, Vienna
- Belgium (4):
  - Centre Hospitalier Universitaire de Liège, Liège, Belgium
  - OLV ziekenhuis Aalst VZW, Aalst
  - Cliniques Universitaires Saint-Luc, Brussels
  - University Hospital Ghent, Ghent
- Germany (15):
  - Evangelisches Herzzentrum Coswig, Coswig
  - Herzchirurgische Klinik Erlangen, Erlangen
  - Universitätsklinikum Essen, Essen
  - Asklepios Kliniken Hamburg GmbH, Hamburg
  - Medizinische Hochschule Hannover, Hanover
  - Universitätsklinikum Heidelberg - Klinik für Herzchirurgie, Heidelberg
  - Universitätsklinikum Schleswig-Holstein, Campus Kiel, Klinik für Herz- und Gefäßchirurgie, Kiel
  - Herzzentrum Leipzig and Helios Health Institute GmbH Leipzig, Leipzig
  - Artemed Klinikum München Süd GmbH & Co. KG, Munich
  - LMU Klinikum Großhadern, Munich
  - Deutsches Herzzentrum München, München
  - Klinikum Nürnberg, Nuremberg
  - Klinikum Oldenburg AöR, Oldenburg
  - Krankenhaus der Barmherzigen Brüder Trier, Trier
  - Universitätsklinikum Ulm, Ulm
- Skåne University Hospital Lund, Lund, Sweden
- Switzerland (3):
  - Hôpitaux Universitaires Genève, Geneva
  - Stadtspital Zürich Clinic for Cardiac Surgery, Zurich
  - Universitätsspital Zürich, Zurich
- United Kingdom (3):
  - Blackpool Teaching Hospitals NHS Foundation Trust/ Blackpool Victoria Hospital, Blackpool
  - Royal Brompton & Harefield Clinical Group (part of Guy's and St Thomas' NHS Foundation TRUST), London
  - Sheffield Teaching Hospitals NHS Foundation Trust, Sheffield

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Schmoeckel M, Thielmann M, Hassan K, Geidel S, Schmitto J, Meyer AL, Vitanova K, Liebold A, Marczin N, Bernardi MH, Tandler R, Lindstedt S, Matejic-Spasic M, Wendt D, Deliargyris EN, Storey RF. Intraoperative haemoadsorption for antithrombotic drug removal during cardiac surgery: initial report of the international safe and timely antithrombotic removal (STAR) registry. J Thromb Thrombolysis. 2024 Aug;57(6):888-897. doi: 10.1007/s11239-024-02996-x. Epub 2024 May 6. PMID 38709456
- [Derived] Schmitto J, De Somer F, Thielmann M, Marczin N, Ruhparwar A, Meyer AL, Hagl C, Matejic-Spasic M, Wendt D, Fan W, Deliargyris EN, Storey RF, Schmoeckel M. Intraoperative antithrombotic drug removal during heart transplantation: A case series from the International Safe and Timely Antithrombotic Removal (STAR) registry. JHLT Open. 2025 Aug 20;10:100369. doi: 10.1016/j.jhlto.2025.100369. eCollection 2025 Nov. PMID 40933270
- [Derived] Storey RF, Hassan K, Meyer AL, Eberle T, deNeve N, Thielmann M, Bernardi MH, Marczin N, Guenther U, Panholzer B, Maechler H, Hunter S, Matejic-Spasic M, Wendt D, Deliargyris EN, Schmoeckel M. Early CABG with intraoperative hemoadsorption in patients on ticagrelor: Real-world data from the international Safe and Timely Antithrombotic Removal (STAR) registry. Cardiovasc Revasc Med. 2026 Jan;82:50-56. doi: 10.1016/j.carrev.2025.02.015. Epub 2025 Feb 28. PMID 40044567
- [Derived] Schmoeckel M, Thielmann M, Vitanova K, Eberle T, Marczin N, Hassan K, Liebold A, Lindstedt S, Machler G, Matejic-Spasic M, Wendt D, Deliargyris EN, Storey RF. Direct-acting oral anticoagulant removal by intraoperative hemoadsorption in CABG and/or single valve surgery: interim analysis of the International Safe and Timely Antithrombotic Removal (STAR) registry. J Cardiothorac Surg. 2025 Jan 20;20(1):74. doi: 10.1186/s13019-024-03326-1. PMID 39833891